CLINICAL TRIAL: NCT04511741
Title: Epidemiological Survey of Children With Prolonged Mechanical Ventilation.
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: CHFudanUCWM
Record Dates: First submitted 2020-08-10; First posted 2020-08-13 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Prolonged Mechanical Ventilation
Keywords: prolonged mechanical ventilation; Children

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- invasive mechanical ventilation
  Interventions: Other: no intervention, it is an observational study.
- non invasive mechanical ventilation
  Interventions: Other: no intervention, it is an observational study.

INTERVENTIONS:
Other: no intervention, it is an observational study. — no intervention, it is an observational study.

SUMMARY:
Mechanical ventilation is an effective treatment for respiratory failure, no more than ten percent of patients with respiratory failure need long-term mechanical ventilation.

DETAILED DESCRIPTION:
Mechanical ventilation is an effective treatment for respiratory failure, no more than ten percent of patients with respiratory failure need long-term mechanical ventilation. There is a lack of data on children with long-term mechanical ventilation in China.The investigators conducted this study to investigate the clinical characteristics of children with long-term mechanical ventilation in China. The investigators conducted a multicenter clinical epidemiological survey.The study included PICU wards in major children's hospitals in China and investigated the causes of prolonged mechanical ventilation, the outcome of long-term mechanical ventilation.PMV definition: continuous invasive or noninvasive ventilation time ≥ 21 days, daily ≥ 6 hours.

ELIGIBILITY:
Inclusion Criteria: patients who need prolonged mechanical ventilation aged from one month to 18 years old.

-

Exclusion Criteria: Other clinical conditions not suitable to participate considered by investigator.

-

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients who need prolonged mechanical ventilation aged from one month to 18 years old.
Sampling Method: Probability Sample
Enrollment: 346 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
the cause of prolonged mechanical ventilation | At enrollment
  This is a categorical variable. The reasons for the prolonged mechanical ventilation wolud be recorded, includes neuromuscular diseases, upper respiratory airway diseases, central nervous system diseases, lower respiratory airway diseases, abnormal ventilation control diseases.

SECONDARY OUTCOMES:
mortality rate | During the procedure (about 2 years)
  The mortality rate among patients received prolonged mechanical ventilation.
the length of prolonged mechanical ventilaton | During the procedure (about 2 years)
  The length of prolonged mechanical ventilaton among patients would be recorded during the hospitalization and after discharging.

CONTACTS AND LOCATIONS:
Overall Officials: Chen Weiming, Study Director — children' hospital of Fudan university
Locations (1):
- Children' hospital of Fudan university, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Racca F, Berta G, Sequi M, Bignamini E, Capello E, Cutrera R, Ottonello G, Ranieri VM, Salvo I, Testa R, Wolfler A, Bonati M; LTV Pediatric Italian Network. Long-term home ventilation of children in Italy: a national survey. Pediatr Pulmonol. 2011 Jun;46(6):566-72. doi: 10.1002/ppul.21401. Epub 2010 Dec 30. PMID 21560263